CLINICAL TRIAL: NCT03963180
Title: Coffee Consumption for Intestinal Function Recovery After Laparoscopic Gynecologic Surgery: a Randomized Controlled Trial
Brief Title: Coffee Consumption for Intestinal Function Recovery After Laparoscopic Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Principal Investigator, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mugla-2
Record Dates: First submitted 2019-05-19; First posted 2019-05-24 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): the control group received 3 cups hot water on the 6th, 12th and 18th hours after the operation
- study group (Experimental): drank 3 cups of caffeinated coffee on the 6th, 12th and 18th hours after the operation.
  Interventions: Other: coffee

INTERVENTIONS:
Other: coffee — All patients were asked to drink the entire 150-mL amounts within 20 minutes under the supervision of a nurse or doctor. Patients were free to drink any amount of water but no more coffee, black tea, or other forms of caffeine, such as soda. Coffee and hot water were prepared with a conventional coffee machine (Nescafe Alegria; 100 g caffeine; Nestlé. Gatwick, United Kingdom).
  Arms: study group

SUMMARY:
Minimally invasive surgery (MIS) has revolutionized women's healthcare. Laparoscopy is an excellent route of MIS. Today, laparoscopic surgery is one of the major procedure in the management of a gynecologic disease. It has revealed benefits of decreased morbidity, earlier discharged, and quicker return to normal daily activities, and shorter hospital when compared to abdominal approach.

Postoperative ileus (POI) defined as an uncomplicated ileus occurring following surgery, resolving spontaneously within 2 to 3 days. Clinically, it is characterized by abdominal distension, a lack of bowel sounds, nausea, vomiting, stomach cramps, and lack of flatus. It leads to morbidity and delays in patient discharge from the hospital, leading to an increased economic burden on the healthcare system. That's why many researchers have focused on the prevent of postoperative ileus; many studies have investigated preventive approaches such as early mobilization of the patient, adequate pain control, epidural anaesthesia, hot pack therapy, motility agents such as metoclopramide, and alvimopan. Although POI incidence has lower after the laparoscopic surgery it remains a major problem during the postoperative period.

Recent studies demonstrated that coffee consumption is associated with improved gastrointestinal function without worsening of postoperative morbidity for both open and laparoscopic surgery. However, until now, no studies investigating the effect of postoperative coffee consumption at laparoscopic gynecologic surgery. Therefore, the investigators performed a randomized controlled trial to assess whether coffee consumption accelerates the recovery of bowel function after laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients underwent total laparoscopic hysterectomy with or without additional surgery *salpingo-oophorectomy,

* salpingectomy,
* pelvic and/or para-aortic lymphadenectomy

Exclusion Criteria:

* patients with hypersensitivity or allergy to caffeine/ coffee,
* patients with thyroid disease,
* patients with inflammatory bowel disease,
* patients with compromised liver function,
* patients with clinically significant cardiac arrhythmia,
* patients with chronic constipation (defined as < 2 bowel movements per week),
* patients with a history of abdominal bowel surgery,
* patients with previous abdominal irradiation,
* the requirement for postoperative care in the intensive care unit >24 hours postoperatively,
* the requirement for nasogastric tube drainage beyond the end of the surgery
* requirement bowel anastomosis
* conversion to laparotomy.

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Time to first passage of flatus | 72 hours
  Patients were checked hourly by auscultation for bowel sounds and were asked to note the time of first flatus and defecation and to inform the observing nurses or assistant.The time to the first passage of flatus after surgery during routine postoperative care.

SECONDARY OUTCOMES:
Time to tolerance of a solid diet | 72 hours
  The time to tolerance of a solid diet was measured from the end of surgery which was defined as when the patients woke up from anesthesia until the patient tolerated the intake of solid food (any food that required chewing) without vomiting or experiencing significant nausea within 4 hours after the meal and without reversion to enteral fluids only
Time to the first bowel movement | 72 hours
  The time to the first bowel movement was defined as the time to the first audible bowel sound during routine postoperative care.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kemal Gungorduk, Muğla
  - Mugla Sıtkı Kocman University Education and Research Hospital, Muğla